CLINICAL TRIAL: NCT01500577
Title: A Randomized Phase II Prevention Trial in Subjects at High Risk for Hormone Non-responsive Breast Cancer
Brief Title: A Prevention Trial in Subjects at High Risk for Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IEO S222/604; 2004-005267-21 (EudraCT Number)
Record Dates: First submitted 2011-12-23; First posted 2011-12-28 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: Prevention; Breast Cancer; Proliferation; Breast Cancer Prevention
MeSH Terms: conditions — Breast Neoplasms | interventions — nimesulide; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nimesulide (Experimental): Nimesulide 100 mg (capsules), 100mg/die every day for 1 year. Oral administration
  Interventions: Drug: nimesulide
- Simvastatin (Experimental): Simvastatin 20 mg (capsules). 20mg/die every day for 1 year. Oral administration
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Placebo (capsules). 1 cps/die every day for 1 year. Oral administration
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: nimesulide — Nimesulide 100 mg (capsules). 100mg/die every day for 1 year. Oral administration
  Other Names: Aulin
  Arms: Nimesulide
Drug: Simvastatin — Simvastatin 20 mg (capsules). 20mg/die every day for 1 year. Oral administration
  Other Names: Sivastin
  Arms: Simvastatin
Other: Placebo — Placebo (capsules). 1 cps/die every day for 1 year. Oral administration
  Arms: Placebo

SUMMARY:
The primary objective of the proposed trial is to assess. The efficacy and the safety of a daily administration of nimesulide or simvastatin to change the expression of a large set of tissue and circulating surrogate endpoint biomarkers (SEBs) of breast carcinogenesis in women at higher risk of developing a hormone non-responsive (ER neg) breast cancer. The primary endpoint is the change in prevalence of atypical cells and cellular proliferation (Ki-67), after 12 months of treatment.

DETAILED DESCRIPTION:
Breast cancer (BC) is one of the four "big killers". The reduction of its incidence and mortality are a top priority. Early diagnosis and screening have modified the average prognosis, nonetheless a significant proportion of BCs ultimately eludes our control. Recently BC prevention has been greatly improved and the chemopreventive efficacy of various compounds, particularly SERMs and more recently AIs (aromatase inhibitors), has been repeatedly documented. However these drugs have shown to be effective almost exclusively in hormone-responsive (ER positive) BCs. At least one-third of BCs will not be influenced by hormonal interventions because of the absence of ER expression since the beginning and another number of cancers will subsequently "escape" the hormonal control and become resistant to tamoxifen and AIs. Unfortunately, ER negativity is frequently combined with other characteristics of biological aggressiveness (high grade and proliferation, overexpression of HER2/neu), resulting in a worse prognosis. Furthermore, women with a family history of breast and ovarian cancer have a higher risk of developing ER negative BC compared with the general population. In particular BRCA-1 mutation carriers have approximately 90% ER negative tumours, and display a characteristic gene expression profile. For all these reasons, methods to better select subjects at higher risk for ER negative BC and strategies to prevent it are actively being sought. Women with BRCA-1 mutations or ERnegative DCIS have a high risk of developing a ER negative tumor. Very importantly, in many of these subjects the onset of BC occurs often early in their lifetime and this one represents not only a clinical, but also a major social issue. Thus, they are suitable candidates for phase II chemoprevention trials with novel agents targeting important molecular pathways. An important potential molecular target for ER negative BC prevention is Cyclo-Oxygenase-2 gene (COX-2) overexpression, which has been strongly correlated with breast carcinogenesis. Other important targets include the inhibition of proteasome and the cholesterol pathway. Agents positively interfering with these pathways, like COX-2 inhibitors and statins, may offer new chances to prevent a form of serious breast disease affecting a large number of subjects worldwide. Importantly, both drugs proposed in this trial add an extensive background of safety to their promising BC prevention effects.

This research is relevant to the following issues in clinical/epidemiological cancer research:

1. the acceptability and the feasibility of cancer chemoprevention in a population at increased risk for breast cancer;
2. the efficacy of the administration of two target-oriented drugs to reduce BC development in a relatively early phase of carcinogenesis;
3. the safety of a low dose of both drugs, with special emphasis to the development of gastrointestinal side effects for nimesulide, and hepatologic side effects for simvastatin;
4. the study of the relationships between tissue biomarkers of carcinogenesis, the presence of intraepithelial neoplasia (including cancer precursors and pre-malignant lesions), and the onset of breast cancer in the placebo arm;
5. the study of the associations between computer-assisted cytometric, morphometric and markovian parameters (nuclear area, DNA index and configurable run length) and the development of breast cancer and their surrogate effect during intervention with nimesulide and simvastatin;
6. the study of the BC associations between insulin-like growth factor-I (IGF-I), IGF binding proteins, hormones and other circulating biomarkers, and the development of breast cancer and their surrogate effect during study intervention.

The proposed study can lead in a 3-year time period to a better understanding of all the above issues. Moreover, we may benefit here of the well-known advantages of the phase II studies on intermediate biomarkers upon larger phase III trials: the combination of lower costs, relatively short times to show results, the possibility to avoid taking "false steps", the concomitant validation of established and novel surrogate biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-65 years old inclusive
* Histologic confirmation of hormone non-responsive DCIS (ER<5%, PgR<5%), or AH or LIN, radically excised in the previous 12 months;
* Positivity for BRCA1 mutation;
* >10% probability of being a BRCA1/2 mutation carrier, according to Berry Parmigiani and/or Couch model;
* Performance Status (SWOG) = 0;
* Unwillingness to be pregnant during the study and three months after drug suspension. Women will be informed that the use of contraceptive pill is contraindicated because it may interfere with the study drugs and may be harmful to a woman who has been diagnosed with breast cancer;
* Willingness to sign the informed consent form

Exclusion Criteria:

* Evidence of residual disease as documented by mammograms, histologic confirmation of margin involvement or distant disease;

  * Previous or concurrent malignancy (with the exception of basal cell carcinoma and CIN);
  * Severe gastrointestinal disorders;
  * Current use of NSAIDs;
  * Current use of statins
  * Current use of fibrates
  * Current use of potent CYP3A4 inhibitors (ciclosporin, mibefradil, itraconazole, ketoconazole, erythromycin, clarithromycin)
  * Proven hypersensitivity to nimesulide and/or simvastatin;
  * Mild or higher alterations of hematologic, liver and renal function (i.e., WBC <3,500/mm3, Plt <120,000/mm3, HgB <10 g/dL, AST >45 U/L, ALT >45 U/L, creatinin >1.5 mg/dL, bilirubin >1.15 mg/dL, CPK 250 mg/dL);
  * CNS diseases and major psychiatric diseases or inability to comply to the protocol procedures;
  * Active infections;
  * Cardiac failure, class I-IV ;
  * Current anticoagulant or antiplatelet aggregation therapy;
  * Mitral and/or tricuspid valvulopathy or valvular prosthesis; Angina; Severe arterial hypertension; Chronic and/or paroxysmal atrial fibrillation; Previous myocardial infarction;
  * Current childbearing and inability to prevent it during the intervention period and for at least 3 months after cessation of treatment;
  * Current lactation.
  * Any other factor that in the investigator's discretion contraindicates the use of one or both drugs.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-04; Primary Completion 2012-11 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Ki 67 variation | baseline and 12 months
  changes of cellular proliferation marker Ki-67 in blood, ductal lavage fluid at the end of treatment withe respect to baseline. A further assessment will be done at the end of a furter 12 months follow-up.

SECONDARY OUTCOMES:
plasma IGF-I, IGFBP-1-2-3, estradiol, estrone sulphate, DHEA-sulphate, SHBG, C-reactive protein, prolactin | 2 years
  change in plasma IGF-I, IGFBP-1-2-3, estradiol, estrone sulphate, DHEA-sulphate, SHBG, C-reactive protein, prolactin at the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Derived] Lazzeroni M, Guerrieri-Gonzaga A, Serrano D, Cazzaniga M, Mora S, Casadio C, Jemos C, Pizzamiglio M, Cortesi L, Radice D, Bonanni B. Breast ductal lavage for biomarker assessment in high risk women: rationale, design and methodology of a randomized phase II clinical trial with nimesulide, simvastatin and placebo. BMC Cancer. 2012 Dec 5;12:575. doi: 10.1186/1471-2407-12-575. PMID 23216985